CLINICAL TRIAL: NCT07391735
Title: Postoperative Pain Procedure Patient Remote Monitoring With MyHealthPal Clinical Study
Brief Title: Post-Surgery Wound Healing Tracking With MyHealthPal App
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Olivia Sutton, Principal Investigator, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025P003153
Record Dates: First submitted 2026-01-28; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Wound Infection and Wound Healing
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MyHealthPal App Users (Experimental): If you choose to be in the app study group, you will be provided with training materials on the MyHealthPal app. After set-up is complete, you will be asked to complete a quick survey on how the set-up went. One day after your surgical procedure (defined as Day 1), you will begin using the MyHealthPal app on your smartphone. For the first 14 days, you will upload a photo of your surgical wound each day and answer a few questions about your wound and how you are feeling. After the first 2 weeks, you will upload a photo of your surgical wound and answer the same questions once every week for 4 months. You will be asked to complete two more surveys regarding your opinion of the app. The app will use your photos and answers to track your wound healing and assess risk of infection. It will use AI to assess risk, and that assessment will be sent to your provider to confirm its accuracy. The app will be used to track your wound healing remotely.
  Interventions: Device: MyHealthPal App
- Controls (No Intervention)

INTERVENTIONS:
Device: MyHealthPal App — MyHealthPal (MHP) is a digital platform for postoperative patients to analyze surgical wound characteristics remotely through photos and additional patient data to provide physicians with SSI risk predictions and inform clinical decision making. It allows postoperative patients to capture and upload wound photos and enter surgery-related medication intake (antibiotics, painkillers), vital signs, wound inputs, and well-being patient data. Patients and providers can access the mobile applications using their own smart devices, while healthcare providers can access the desktop portal through a personal computer. MHP provides a prediction report for healthcare providers anytime a patient enters any data. If the patient uploads a high quality surgical incision photo, MHP's prediction reports include an SSI risk prediction: elevated risk or standard risk. MHP's AI-based algorithm analyzes wound photos for characteristics indicative of infection and provides risk predictions for providers.
  Arms: MyHealthPal App Users

SUMMARY:
We want to explore the use of a smartphone app that allows patients to take photos of their wounds in early stages of healing, so that clinicians can monitor wound-healing remotely with the assistance of an AI program.

Participants will choose whether they want to be in the control group or the app group. People in the app group will be asked to download an app on their personal smartphone before their surgery. After the procedure, participants will upload a photo of their surgery site as well as answer some questions about its characteristics either on a daily or weekly basis. A healthcare provider and the app's AI algorithm will observe this information to determine the risk of infection. People in the control group will not be asked to use the app. Their medical record will be monitored by study staff intermittently to see if they develop infection. This study will take approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years old and older).
* Ability to understand consent process and questionnaires. Patients with ready access to a smartphone, compatible smart device (operating system 5.0 version, also known as Lollipop, for Android and 13 or later version for iOS), smartphone aptitude, smartphone with sufficient memory space for the relevant app, and willingness to participate in the study as assessed by a questionnaire.
* Patients undergoing one of the following surgeries within the Brigham and Women's Pain Management Practice:

  1. Spinal cord stimulator implantation
  2. Spinal cord stimulator explant
  3. Spinal cord stimulator revision
  4. Intrathecal pump implantation
  5. Intrathecal pump explant
  6. Intrathecal pump revision
* Ability to attend all standard surgery follow-up appointments at Brigham and Women's Hospital.
* Ability to understand and sign written informed consent documents.

Exclusion Criteria:

* Cognitive or physical impairment that would prevent patient from entering data in MHP.
* Any acute or chronic condition that would limit the ability of the patient to participate in the study.
* Any patient who is experiencing an ongoing infection prior to undergoing a surgical revision/explant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Imageability | From enrollment to end of app usage at 16 weeks post-surgery
  Imageability is defined as the percentage of wound incision photos that received an SSI risk prediction (high enough quality photos) by MHP's artificial intelligence algorithm among all photos uploaded by patients. High imageability is a critical step in MHP's predictive effectiveness. MHP Patient app guides patients on how to take surgical incision photos that are high enough quality for analysis. Target imageability percentage is greater than or equal to 95%.
Positive/negative percent agreement | From enrollment to end of app usage at 16 weeks post-surgery
  Positive/negative percent agreement will be sought for each MHP prediction by receiving feedback from one of the study investigators. The investigator will be prompted to agree or disagree with each MHP prediction (elevated or standard risk for an SSI). Final positive/negative agreement percentage will be calculated after the last subject completes the 16-week study period.
Patient Usage/Data Entry | From enrollment to end of app usage at 16 weeks post-surgery
  MHP effectiveness is directly dependent on patient use and data entry. This study aims to demonstrate >70% patient compliance with the monitoring plan data entry requirements. Patient compliance with data entry will be calculated by input category, wound photo, wound inputs, vital signs, medication adherence, and well-being, as well as overall patient compliance with all data entry requirements that are defined in the patient monitoring plan.

SECONDARY OUTCOMES:
Clinician Feedback | From first enrollment to final subject's end of app usage at 16 weeks
  When clinicians agree or disagree with MHP's prediction, they are encouraged to submit their feedback on incision characteristics that they observe in the photos. This feedback is particularly helpful in identifying early/leading indicators of SSIs. In this study, a secondary objective is for clinicians to submit their comments greater than or equal to 95% of the time they have agreed or disagreed with a prediction.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia M Sutton, MD, Principal Investigator — Brigham and Women's Anesthesiology Department